CLINICAL TRIAL: NCT06857123
Title: Mechanical and Molecular Determinants of Cartilage Response to Exercise
Brief Title: Feasibility of Resting Intervals During Exercise Programs for Individuals With Knee Osteoarthritis
Acronym: CaRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Sara R. Piva, Professor and Vice Chair for Research, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23050179
Record Dates: First submitted 2025-01-17; First posted 2025-03-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthristis
Keywords: Knee; Osteoarthritis; exercise; feasibility
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise With Rest (Experimental): Participants in this arm exercise 3 times a week for 12 weeks. Exercise program consists of warm-up, strengthening exercises of the lower major extremity muscle groups, and aerobic training using a treadmill. These sessions include two 45 minute rest periods between exercises and take about two and a half hours.
  Interventions: Behavioral: Exercise with Rest
- Exercise Without Rest (Active Comparator): Exercise without Rest
  Interventions: Behavioral: Exercise without Rest

INTERVENTIONS:
Behavioral: Exercise with Rest — Participants in this arm exercise 3 times a week for 12 weeks. Exercise program consists of warm-up, strengthening exercises of the lower major extremity muscle groups, and aerobic training using a treadmill. These sessions include two 45 minute rest periods between exercises and take about two and a half hours.
  Arms: Exercise With Rest
Behavioral: Exercise without Rest — Participants in this arm exercise 3 times a week for 12 weeks. Exercise program consists of warm-up, strengthening exercises of the lower major extremity muscle groups, and aerobic training using a treadmill. These sessions include minimal resting periods between exercises and take about one hour.
  Arms: Exercise Without Rest

SUMMARY:
This pilot randomize trial tests the feasibility of administering two different exercise programs in people with knee osteoarthritis. One group receives the exercise program administered as usual, and the other group received the exercise program with resting intervals.

DETAILED DESCRIPTION:
Participants will be randomly assigned to 1 of 2 treatment groups. Both groups do the same exercise program 3 times a week for 12 weeks on nonconsecutive days. The only difference is that one group will perform the exercises with small resting periods between exercises as normally done in clinical practice. The other group will have two long rests of 45 minutes during the exercise training session. Before and after the exercise programs, participants will undergo a series of assessments including gait analysis, MRI imaging of knees, tests of muscle strength and physical performance. Questionnaires will be completed. Blood and synovial fluid will be collected as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 79 yo.
* Clinical diagnosis of primary, early to moderate stage knee osteoarthritis.
* BMI range < 35 kg/m2.
* Sedentary lifestyle
* Knee joint is the most painful joint in the body.
* Ability to speak and understand English.
* Willingness to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Non-OA disease of the knee.
* Advanced knee osteoarthritis
* Knee injection in the past 3 months.
* Major knee trauma/surgery in the past 5 years or previous knee surgery with hardware limiting cartilage assessment..
* Participate in regular exercise or physical activity .
* Participation in an intervention study for knee OA.
* Currently using a cane, walker or crutches to walk.
* History of cardiovascular disease or hypertension not controlled by medication.
* Two or more unexplained falls in the past year.
* Inflammatory, autoimmune disorders, neurological, systemic, muscular, or connective tissue conditions that affect walking or ability to exercise.
* Contraindication to MRI.
* Medical condition or characteristic of the participant that could place the individual at increased risk or preclude s/he from complying with study procedures.
* Pregnant female.
* Acute or terminal illness.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | The time frame for this outcome is from the enrollment period up to randomization. This outcome measure is independent of treatment assignment.
  The number of eligible individuals who are randomized out of all eligible individuals.

SECONDARY OUTCOMES:
Safety of interventions | 3 months (window of 1 month)
  The number of adverse events related to study participation in each arm

OTHER OUTCOMES:
Adherence to Intervention | 3 months (window of 1 month)
  The number of intervention sessions attended out of the total number of intervention sessions prescribed in the study.
Study retention | 3 months (window of 1 month)
  The number of participants in each intervention arm who attend the follow-up assessment visit out of the number of participants randomized to each intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Piva, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the conclusions of this study will be available upon request to the principal investigators. The data will include participants demographic and biomedical information, along with primary and secondary outcome measures. The data dictionary will be provided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available at the time of the publication of the pilot feasibility results in peer-reviewed medical journal.
Access Criteria: IPD will be available upon request to the principal investigators. The data will include participants demographic and biomedical information, along with primary and secondary outcome measures. The data dictionary will be provided. Non-identifiable data will be shared in CSV files.